CLINICAL TRIAL: NCT06603181
Title: Effect of Extracorporeal Shock Wave Therapy (ESWT) and Phonophoresis Treatment on Pain, Function, Grip Strength and Tendon Thickness in Ultrasonography in Patients With Lateral Epicondylitis.
Brief Title: Effect of Extracorporeal Shock Wave Therapy (ESWT) and Phonophoresis Treatment in Patients With Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Nazife Kapan, Asst. Prof., Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AEÜ-NK-LE
Record Dates: First submitted 2024-05-07; First posted 2024-09-19 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2024-09

CONDITIONS: Lateral Epicondylitis; Extracorporeal Shock Wave Therapy; Phonophoresis
MeSH Terms: conditions — Tennis Elbow | interventions — Phonophoresis; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Conventional Treatment Patients in this group will be given activity modification and home exercise program training, including stretching and eccentric strengthening exercises. Patients will be asked to perform the exercise treatment in 3 sets of 10 repetitions. Additionally, a splint will be recommended to rest the arm.
  Interventions: Other: conventional treatment
- GroupB (Experimental): Conventional Treatment and Phonophoresis Patients in this group will receive phonophoresis treatment in addition to a home exercise program and splint. A US device (Intelect 2776 Combo; Chattanoga Group, Inc, Chattanoga, TN) will be used for phonophoresis. The gel containing 10% naproxen will be mixed with aquasonic us gel to better deliver the drug through the body. Continuous mode at 1watt/cm2 1mhz frequency will be applied around the lateral epicondyle for 5 minutes. Sessions will be applied 5 sessions per week for 2 weeks.
  Interventions: Other: conventional treatment; Other: phonophoresis
- Group C (Experimental): Conventional Treatment and Ekstrakorporeal shock wave therapy Patients in this group will receive ESWT treatment in addition to a home exercise program and splint. ESWT; With the MODUS ESWT system, 2 sessions per week will be applied to the lateral epicondyle (2.4 bar intensity, 15 Hz frequency, 1500 pulses) for 2 weeks (Modus ESWT® RadialShockwaveTherapy).
  Interventions: Other: conventional treatment; Other: extracorporeal shock wave therapy

INTERVENTIONS:
Other: conventional treatment — exercise and splint
Other: phonophoresis — exercise, splint and phonophoresis
  Arms: GroupB
Other: extracorporeal shock wave therapy — exercise, splint and ESWT
  Arms: Group C

SUMMARY:
This study aimed to investigate the effects of Extracorporeal Shock Wave Therapy and phonophoresis treatment on pain, function, hand grip strength and tendon thickness in ultrasonography in patients with lateral epicondylitis.

DETAILED DESCRIPTION:
Lateral epicondylitis (LE) is tendinopathy of the forearm extensor muscles, often caused by overuse or repetitive use, forced wrist extension, or direct trauma to the epicondyle. It is the most common cause of lateral elbow pain. Although also known as tennis elbow, lateral epicondylitis often develops as a work-related condition and is therefore a significant public health problem.

ESWT; It involves transmitting high-intensity acoustic pressure waves produced by electrohydraulic, electromagnetic or piezoelectric devices to the target area of the body in a short time through the gel. It has been reported that ESWT increases collagen synthesis in tendons, bones and other soft tissues, accelerates vascularization and reduces pain.

ultrasound; It has been used for many years in the treatment of musculoskeletal disorders such as tendinitis, epicondylitis, tenosynovitis, bursitis and osteoarthritis. It produces acoustic waves through the conversion of electrical energy. These waves turn into heat as they pass through tissues at different resistance levels. Ultrasound is also used to enhance percutaneous absorption of drugs in phonophoresis applications.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65
* Those who signed the informed consent form
* Painful palpation of the lateral epicondyle
* Positive Mill's, Maudsley's and Cozen's tests
* Patients who have had complaints for at least 3 months

Exclusion Criteria:

* Those who have had corticosteroid, PRP, prolotherapy, hyaluronic acid etc. injections into the elbow area within 3 months or those who have received physical therapy
* Those with cervical radiculopathy
* Those who have had surgery on the elbow
* Those with an open wound on the elbow
* Those with a history of malignancy
* Those with rheumatological diseases
* Those with neurological diseases
* Pregnancy
* Infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | baseline, 2th week, 12th week
  VAS is a pain rating scale with numbers 0 and 10. Here 0 means 'no pain' and 10 means 'unbearable pain'. The participant will rate the pain according to the scale. Patients' night, rest and activity pain will be evaluated separately.
Patient-based lateral epicondylitis assessment questionnaire | baseline, 2th week, 12th week
  It is a specific assessment questionnaire for lateral epicondylitis. It consists of two parts. In the first part, the pain in the affected arm is evaluated, and in the second part, the level of functionality is evaluated. In the second part, the functionality level is divided into two parts: specific activities and daily activities. In total, the best score is evaluated as 0 and the worst score is evaluated as 100.

SECONDARY OUTCOMES:
Quick-DASH | baseline, 2th week, 12th week
  It is an evaluation questionnaire that measures activity and participation limitations in all upper extremity disorders. In the survey, patients' difficulties during daily living activities are questioned with 11 questions. Each answer is scored on a Likert scale from 1 to 5, from best to worst.
hand grip strength | baseline, 2th week, 12th week
  It will be done with a Jamar dynamometer. Patients will be seated in a chair with their elbows flexed at 90 degrees and their forearms in a neutral position. They will be asked to squeeze the dynamometer for a maximum of 3 seconds, and this will be repeated 3 times, with a 60-second rest in the meantime. The average of 3 results will be recorded.
tendon thickness | baseline, 2th week, 12th week
  Extensor tendon thickness measurement will be performed by the same researcher under clinical ultrasound guidance. Plato technique will be used. The plateau is located between the attachment site of the extensor tendon and the humeroradial joint. Tendon thickness is measured perpendicularly from the plateau to the tendon surface.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran University, Kırşehir, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided